CLINICAL TRIAL: NCT06632639
Title: Effect of Lateral Wedged Insoles With Subtalar Strapping on Genu Varum With Medial Compartment Knee Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Abdelmoniem Ali Hassanien, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005074
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Genu Varum
MeSH Terms: conditions — Genu Varum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corrective exercise protocol + Lateral wedged insoles with subtalar strapping (Experimental): They will receive the corrective exercise protocol in addition to the lateral wedged insoles with subtalar strapping for 12 weeks.
  Interventions: Other: Corrective exercise protocol; Other: Lateral wedged insoles with subtalar strapping
- Corrective exercise protocol (Active Comparator): They will receive the same corrective exercise protocol alone for 12 weeks.
  Interventions: Other: Corrective exercise protocol

INTERVENTIONS:
Other: Corrective exercise protocol — The program requires 60 minutes consisting of a ten-minute warm-up, a forty-minute Thera-band exercise, and a ten-minute cool-down. Thera-band exercises are to improve the external rotators, and the extensors and for strengthening the quadriceps and the gluteus. A set consists of 15 reps, each of the exercise methods consisted of three sets.
Other: Lateral wedged insoles with subtalar strapping — A silicon rubber 10 mm lateral wedge has a 10 mm lateral elevation and a 75 mm width, which has an approximately 7.6 inclination. This silicon rubber material is usually used for cosmetic remodeling and has a natural form-fit to the skin. The 75 mm width silicon rubber is scaphoid shaped and it is suitable for attachment to a barefoot of all of the subjects. The rational for using this inclination is that 7.6 is approximately the median between 5 and 10. Patients will be instructed to use the wedge in an appropriate shoe (not high heels or narrow-toed shoes), 1 h a day during the first week. The duration of use gradually will be increased to the minimum of 8 h a day.
  Arms: Corrective exercise protocol + Lateral wedged insoles with subtalar strapping

SUMMARY:
The purpose of the study is to investigate the effect of lateral wedged insoles with subtalar strapping in genu varum with medial compartment knee pain on:

1. Space between knees (measured by vernier calipers)
2. Degree of genu varum deformity (Femorotibial angle (FTA)) measured on long film weight bearing x-ray)
3. Pain level (Measured by VAS)
4. Hind foot angle (measured by long axial hindfoot alignment view)
5. Functional outcome (measured by the lower extremity function scale)
6. Functional performance (measured by the 6 minute walk test)

DETAILED DESCRIPTION:
Genu varum is known as one of the most common lower limb abnormalities. Genu varum is reported to occur 15 to 20% in the whole population. In most cases, this deformity occurs between tillage damage and degeneration in the medial compartment of the knee joint in the long term, because of the imposed imbalanced force on medial and lateral compartments of knees.

Incidence of rachitic genu varum in preschool children: A more recent study from 2016 estimated the incidence of vitamin D deficient rachitic genu varum among preschool children in Egypt, finding it to be 13.1% of all children's orthopaedic diseases at the National Institute of Neuromotor System.

Prevalence of lower limb deformities in primary school students: A 2021 study reported a much lower prevalence of genu varum (0.09%) among primary school students in Egypt. This suggests that the condition may be more prevalent in younger children and decrease in severity with age.

Surgical treatments, such as high tibial osteotomy and total knee arthroplasty (TKA) have been performed. Although this type of surgery has provided successful clinical results, it is often costly for the patients and it forces them to get over complications. In particular, more than 500,000 cases of TKA are annually performed in the US, and approximately three billion dollars are spent on TKA. Alternatives to surgical treatment are required to lighten the patient's burden and the medical costs.

lateral wedged insole significantly reduces the knee varus moment during walking compared to the barefoot condition with no insole. In particular, the strapping insole reduces the varus moment more than the lateral wedged insole alone in moderate OA.

Exercises of correcting genu varum might have positive effects on changes in hip joint angle, Q angle, and knee space distance, and lower limb deformity not by structural causes but by muscular imbalance might be corrected via consistent exercises.

The results of this study could potentially inform the treatment approach for individuals with medial compartment knee pain caused by genu varum. Also provides a non-invasive and cost-effective alternative to managing knee pain, which can improve the quality of life for individuals suffering from this condition. Additionally, this study adds to the body of knowledge on the effectiveness of corrective orthoses in managing musculoskeletal disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aged 20-60.
* Patients with medial compartment pain. Pain level of 3 or more on the VAS.
* Patients with varus deformity are defined as those Those whose femorotibial angle measures 5-10 degrees of genu varum on long film weight bearing x-ray.
* Patients with grade one O.A. on Kellgren-Lawrence classification system or without O.A.
* BMI less than 35
* Patients with decompensated hind foot (hind foot varus)

Exclusion Criteria:

* Patients already wearing custom wedged insoles.
* Patients with other inflammatory conditions like rheumatoid arthritis or systematic inflammatory arthritis.
* Patients with central or peripheral nervous system disease.
* Any previous surgical procedure to the knee joint.
* Patients who are unable to walk without assistance (cane or a walker).
* Pregnancy
* Uncooperative patient types due to mental disorders or others.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-10-12 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Distance between knees using vernier calipers | 12 weeks
  To measure the distance between the participants' knees, we have them put both feet together, so that both malleolus bones were together, and measured the space between the tibia and medial condyle using vernier calipers.

SECONDARY OUTCOMES:
Degree of genu varum deformity measured by long film weight bearing X-Ray | 12 weeks
  The femorotibial angle in the frontal plane is the angle formed by the intersection of anatomical axes of the femur and tibia. In normal knee alignment, there is an approximately 5°-7° valgus femorotibial angle.
Pain level measured by the visual analogue scale (VAS) | 12 weeks
  The VAS is a uni-dimensional measure of pain intensity.It is a continuous scale that comprises of a horizontal line of 10 cm in length. The scale is anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 10). A higher score indicates greater pain intensity.
Hind foot angle measured by long axial hindfoot alignment view | 12 weeks
  The film cassette is lying on the floor and the subject is standing on the film cassette. The inclination angle of the beam is 45° to the floor.
Functional outcome measured by lower extremity function scale (LEFS) | 12 weeks
  The lower extremity function scale (LEFS) is a region specific outcome measure that was designed to assess activity limitations due to musculoskeletal disorders of the lower extremity. LEFS has 20 items each scored on 0-4 Likert scale and the overall score on the scale is produced by summing scores on all items. LEFS score range from 0 to 80 with higher score indicating better functional ability.
Functional performance measured by the 6 minute walk test | 12 weeks
  The patients will walk as far a distance as possible within 6 minutes. They will be instructed to walk as fast as possible, but running or jogging will not be allowed. Standardized encouragement and updates on the remaining time for the 6MWT will be provided at each minute mark. When the patient turns around a cone (set 30 meters away), it will be marked on a worksheet. After 6 minutes, the patients will be told to stop immediately, and a small piece of tape will be placed just in front of their shoes. The additional distance covered (in the final 30-meter stretch) will be measured to the nearest centimeter. Finally, the total distance walked by each patient in 6 minutes will be calculated and recorded. Patients will be permitted to rest by standing or leaning against the wall during the test trial, but the timer will continue to run.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Abdulrahman, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Faculty of physical therapy, Cairo University, Giza, Egypt